CLINICAL TRIAL: NCT02268695
Title: TPExtreme: Randomized, Controlled Trial of Platinum-Cetuximab Combined Either With Docetaxel (TPEx) or With 5FU (Extreme) in Patients With Recurrent/Metastatic Squamous Cell Cancer of the Head and Neck
Brief Title: Platinum-Cetuximab Combined With Docetaxel or With 5FU in Patients With Recurrent/Metastatic HNSCC
Acronym: TPExtreme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other); AIO-Studien-gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2014-01
Record Dates: First submitted 2014-10-13; First posted 2014-10-20 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Recurrent/Metastatic HNSCC; Taxanes
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; Docetaxel; Cetuximab; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EXTREME: Cisplatin, 5-FU and Cetuximab (Active Comparator): Chemotherapy: 6 cycles (every 3 weeks) of Cisplatin (100 mg/m² iv on Day1), 5FU (4000 mg/m² total dose starting on day 1 and during 96h in continuous infusion), and Cetuximab (loading dose of 400 mg/m² iv on Day1, then 250 mg/m² iv weekly).
  If cisplatin is not tolerated and/or when the total cumulative dose of cisplatin (including prior administration) reaches 600 mg/m², cisplatin has to be replaced by carboplatin, AUC 5 (but not exceeding 750 mg), except in the case of bleeding tumor.
  Cetuximab maintenance : cetuximab continuation (250 mg/m² iv weekly) will begin only if at least disease stabilization is observed at the end of chemotherapy, and will be continued until PD or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: 5-Fluorouracile; Drug: Cetuximab
- TPEx: Cisplatin, Docetaxel and Cetuximab (Experimental): Chemotherapy: 4 cycles (every 3 weeks) of Cisplatin (75 mg/m² iv on Day1), Docetaxel (75 mg/m² iv on Day1), and Cetuximab (loading dose of 400 mg/m² iv on Day1, then 250 mg/m² iv weekly).
  If Cisplatin is not tolerated, cisplatin is replaced by carboplatin, AUC 5 (but not exceeding 750 mg), except in the case of bleeding tumor.
  Primary prophylactic administration of GCSF must be administered systematically after each cycle of chemotherapy.
  Cetuximab maintenance : cetuximab continuation (500 mg/m² iv every two weeks) will begin only if at least disease stabilization is observed at the end of chemotherapy, and will be continued until PD or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Cetuximab; Drug: granulocyte colony-stimulating factor (G-CSF)

INTERVENTIONS:
Drug: Cisplatin
Drug: 5-Fluorouracile
  Arms: EXTREME: Cisplatin, 5-FU and Cetuximab
Drug: Docetaxel
  Arms: TPEx: Cisplatin, Docetaxel and Cetuximab
Drug: Cetuximab
Drug: granulocyte colony-stimulating factor (G-CSF)
  Arms: TPEx: Cisplatin, Docetaxel and Cetuximab

SUMMARY:
This study evaluates the efficacy of the new docetaxel-cisplatin-cetuximab regimen (TPEx) versus the standard platinum-5FU-cetuximab EXTREME regimen as a first-line treatment in recurrent and/or metastatic HNSCC. Half of patients will be treated by TPEx regimen, while the other half will be treated by EXTREME regimen.

DETAILED DESCRIPTION:
The EXTREME regimen, i.e. cetuximab added to platinum (100 mg/m² every 3 weeks ) and 5FU (96h continuous infusion at 1000 mg/m²/day every 3 weeks) during 6 cycles of treatment and continued as maintenance in patients with stable disease, is currently the standard of care in first line recurrent metastatic HNSCC.

From our previous experience (phase II GORTEC "TPEx" study), the TPEx regimen of 4 cycles of docetaxel-cisplatin-cetuximab followed by maintenance with cetuximab every 2 weeks seems more efficient (overall survival) compared to EXTREME regiment. Docetaxel combined with cisplatine (each administered at 75mg/m² every 3 weeks) also appeared more convenient than the standard Cisplatin-5FU-Cetuximab EXTREME regimen (4 cycles of chemotherapy instead of 6 cycles and no i.v. continuous infusion). Toxicity was manageable with G-CSF support. In addition the toxicity / efficacy profile also seems favourable as suggested by the excellent dose intensity achieved and the high rate of patients (78%) who were able to start maintenance therapy.

Taking together all these considerations, the TPEx regimen might be a good substitute for EXTREME as first-line treatment in patients with recurrent metastatic HNSCC, and it is justified and necessary to perform a direct comparison in a randomized trial to further test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis squamous cell carcinoma of head and neck: oral cavity, oropharynx, hypopharynx, larynx (histological confirmation is mandatory at least for initial diagnosis)
* Recurrence and/or metastatic disease not suitable for local therapy
* At least one measurable lesion (RECIST) by CT or MRI
* PS < 2
* Age ≥ 18 years and < 71 years
* Clearance of creatinine > 60ml/mn (MDRD)
* Haematological function as follows: absolute neutrophil count > 1.5 x 109/l, platelet > 100 x 109/l, hemoglobin ≥ 9.5 g/dl
* Hepatic function as followed: bilirubin ≤ Upper limit of normal (ULN); SGOT/SGPT < 1.5 ULN; AP < 2.5 ULN
* Estimated life expectancy > 12 weeks
* Informed Consent Form signed
* Affiliation to an health insurance
* Negative pregnancy test in women of childbearing potential within 14 days prior to treatment initiation (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilization). Both men and women (of childbearing potential) who are sexually active must use adequate contraception, during and for at least 6 months post-treatment.

Exclusion Criteria:

* Patients with nasopharyngeal cancer, paranasal sinus cancer or unknown primary
* Prior systemic chemotherapy for the head and neck carcinoma, except if given as part of a multimodal treatment for locally advanced disease which was completed more than 6 months prior to study entry
* Surgery (excluding diagnostic biopsy) or radiotherapy within 6 weeks before study entry
* Contra-indication to receive cisplatin
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Administration of prophylactic phenytoin
* Recent or planed yellow fever vaccination
* Prior dose of cisplatin > 300 mg/m² (a patient who received prior RT + 3 cycles of cisplatin or 3 cycles induction TPF, i.e. total dose of cisplatin ≤ 300 mg/m², for locally advanced primary HN cancer can be included)
* Prior anti-EGFR treatment received less than 12 months before enrolment in the trial
* Known hypersensitivity reaction to 5FU, cisplatin, carboplatin, docetaxel or cetuximab
* Documented or symptomatic brain or leptomeningeal metastasis
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months
* Malignancies within 5 years prior to randomization, with the exception of adequately treated basal or squamous cell skin cancer and carcinoma in situ of the cervix
* Active infection (infection requiring IV antibiotics), including active tuberculosis and known and declared human immunodeficiency virus (HIV).
* Significant disease which, in the judgment of the investigator, would make the patient inappropriate for entry into the trial.
* Any social, personal, medical and/or psychologic factor(s) that could interfere with the observance of the patient to the protocol and/or the follow-up and/or the signature of the informed consent.
* Pregnant or breast feeding women

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | Until patient death or at least one year after the end of the treatment
  Overall survival is defined as the time to death from any cause measured from randomization. Patients with disease progression may be treated with off protocol therapy but will be followed for overall survival evaluation.

SECONDARY OUTCOMES:
Objective response rate | At 12 weeks
  Objective response rate (complete response (CR) or partial response (PR) according to RECIST 1.1 criteria and assessed by central imaging review) at 12 weeks. For the statistical analysis patients not evaluable (whatever the reason, including death) will be considered as failure (i.e. no CR, no PR).
Best overall tumor response rate | until progression or at least one year after the end of the treatment
  Best overall tumor response rate (RECIST 1.1 criteria) during chemotherapy and maintenance: CR or PR or SD confirmed for CR or PR by a second assessment 6 weeks later
Progression free survival | until progression or death or at least one year after the end of the treatment
  Progression free survival (PFS): minimum time from randomization to progression as defined by RECIST 1.1 criteria or to death from any cause. Patients who don't have any of these events are censored at the date of last follow-up.
Time to Progression | until progression or death or at least one year after the end of the treatment
  Time to Progression (TTP): minimum time from randomization to progression as defined by RECIST 1.1 criteria. In case of death from other cause than cancer and no prior progression, the patient will be censored at the time of death. In case of death related to cancer without an accurate date of progression before death, the patient will be considered in progression at the time of death. In the event of no progression and no death, the patient will be censored at the date of last follow-up.
Toxicity | until the end of the maintenance, an expected average of 4 months of maintenance
  Toxicity (according to CTC-NCI V4): all grades
Compliance | until the end of the maintenance, an expected average of 4 months of maintenance
  Compliance: Insufficient compliance for cetuximab is defined as a patient missing more than 2 consecutive infusions of cetuximab, even if the missed infusions are due to toxicity. Insufficient compliance for chemotherapy is defined as a patient missing more than 2 consecutive infusions of chemotherapy, even if the missed infusions are due to toxicity.
EORTC QLQ-C30 | At baseline before treatment, at Week 12, Week 18 and at Week 26
  Health related quality of life (QoL) assessed by EORTC QLQ-C30. The primary endpoint of the QoL study is the global health status/quality of-life scale of the QLQ-C30 questionnaire
EuroQol-5D | At baseline before treatment, at Week 12, at Week 26 and then every 2 months.until death or at least one year after the end of the treatment
  Quality-adjusted life-years (QALYs) based on Euroqol EQ-5D measurements
Net monetary benefit | until death or at least one year after the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joel GUIGAY, MD, Study Chair — Centre Antoine Lacassagne, Nice, France; Jean BOURHIS, MD, PhD, Study Director — GORTEC President; Ricardo MESIA, MD, Principal Investigator — Instituto Catalá de Oncologia (ICO), Barcelona, Spain; Ulrich KEILHOLZ, MD, Principal Investigator — Charité Campus Benjamin Franklin, Berlin, Germany
Locations (17):
- France (15):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de la Dracénie, Draguignan
  - Centre Médical de Forcilles, Férolles-Attilly
  - Clinique des Ormeaux, Le Havre
  - Centre Hospitalier de Bretagne Sud (CHBS), Lorient
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - ICM Val d'Aurelle, Montpellier, Montpellier
  - Centre Antoine-Lacassagne, Nice
  - Val de Grace, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de l'Ouest (ICO) René Gauducheau, Saint-Herblain
  - L'Institut de Cancérologie de Lorraine (ICL) Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Charité Campus Benjamin Franklin, Berlin, Germany
- Instituto Catalá de Oncologia (ICO), Barcelona, Spain

REFERENCES:
- [Derived] Atsou K, Auperin A, Guigay J, Salas S, Benzekry S. Mechanistic Learning for Predicting Survival Outcomes in Head and Neck Squamous Cell Carcinoma. CPT Pharmacometrics Syst Pharmacol. 2025 Mar;14(3):540-550. doi: 10.1002/psp4.13294. Epub 2024 Dec 25. PMID 39722558
- [Derived] Guigay J, Auperin A, Fayette J, Saada-Bouzid E, Lafond C, Taberna M, Geoffrois L, Martin L, Capitain O, Cupissol D, Castanie H, Vansteene D, Schafhausen P, Johnson A, Even C, Sire C, Duplomb S, Evrard C, Delord JP, Laguerre B, Zanetta S, Chevassus-Clement C, Fraslin A, Louat F, Sinigaglia L, Keilholz U, Bourhis J, Mesia R; GORTEC; AIO; TTCC, and UniCancer Head and Neck groups. Cetuximab, docetaxel, and cisplatin versus platinum, fluorouracil, and cetuximab as first-line treatment in patients with recurrent or metastatic head and neck squamous-cell carcinoma (GORTEC 2014-01 TPExtreme): a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2021 Apr;22(4):463-475. doi: 10.1016/S1470-2045(20)30755-5. Epub 2021 Mar 5. PMID 33684370